EFFICACY AND NEURAL MEDIATORS OF RESPONSE TO TRAUMA MANAGEMENT THERAPY FOR PTSD NCT03449576 Analysis of primary clinical outcome hypothesis for D2354-R "Efficacy and Neural Mediators of Response to Trauma Management Therapy for PTSD"

A regression approach was used to test the effect of treatment type (TMT, EXP+EDU) on both primary (CAPS-5 and SAS-SR) and secondary (PCL-5, AQ, ITS) outcome measures across Time (pre-treatment, post-treatment). The Time x Treatment interaction was be used to test whether TMT improves outcomes relative to EXP+EDU, and age was entered as a co-variate as the two treatment arms differed in age at baseline.